CLINICAL TRIAL: NCT01551524
Title: A Dose Escalation Phase I Study of Asparec®(mPEG-R-Crisantaspase) Administered as Intravenous (IV) Infusion in Patients With Relapsed or Refractory Hematological Malignancies
Brief Title: Phase I Study of mPEG-R-Crisantaspase Given IV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: EUSA SAS (Unknown); The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZPO2-CLT-001; 2011-000295-34 (EudraCT Number)
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-02

CONDITIONS: Hematologic Malignancies
Keywords: Leukemia; Lymphoma; C240588.448; C115.378.400
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravenous Erwinia (Experimental)
  Interventions: Biological: mPEG-r-crisantaspase

INTERVENTIONS:
Biological: mPEG-r-crisantaspase — IV infusion over 60 minutes of mPEG-r-crisantaspase given once every two or four weeks for two administrations. Based on non-clinical data, 500IU/m2 has been selected as the starting dose. Dose selection will proceed based upon safety and pharmacokinetic data but escalation will not exceed 100%
  Other Names: Asparec

SUMMARY:
This study is an open label, multicenter study with a dose escalation of Asparec® administered once every two to four weeks for two administrations. The primary objective of this study is to determine the Maximum Tolerated Dose following one single dose of Asparec when administered in a population of patients with relapsed or refractory hematological malignancies, as measured by Dose Limiting toxicities. There are secondary objectives which are to evaluate the safety of Asparec and to determine the PK profile as assessed by measurement of plasma L-asparaginase enzymatic activity following single and repeated doses of Asparec. Patients response rate will be evaluated and Anti-Asparec antibodies will be measured.

DETAILED DESCRIPTION:
Planned sample size: Up to 36 evaluable subjects will be enrolled in the study: a maximum of 30 subjects for the dose escalation phase and up to a maximum of 12 patients in the expansion phase.

Inclusion criteria consists of:

Patients with any relapsed or refractory hematological malignancy, for which standard curative or life prolonging treatment does not exist, or is no longer effective or tolerable.

For the following hematological malignancies, patients must have received at least: Low rade NHL: 3 prior lines of therapy, ALL, aggressive NHL and other hematological malignancies: 2 prior lines of therapy, Aged 18 to 50 years and ECOG performance status of 1, 1 or 2.

All patients will be treated with Asparec once every two to four weeks for two IV administrations infused in 60 minutes. Patients without Disease Progression may receive additional administrations, each administration starting at least 14 days but no later than 28 days after the previous Asparec administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any relapsed or refractory hematological malignancy, for which standard curative or life prolonging treatment does not exist, or is no longer effective or tolerable.
* For the following hematological malignancies, patients must have received at least:

  * Low grade NHL:

    * 3 prior lines of therapy and ALL,
  * aggressive NHL and other hematological malignancies:

    * 2 prior lines of therapy.
* Ages 18 to 50 years and
* ECOG performance status of 0, 1 or 2,
* ability to understand and to sign a written informed consent and
* have a life expectancy of greater than or equal to 90 days

Exclusion Criteria:

* Any active CNS disease,
* previous greater than or equal to grade 3 allergic reaction to Erwinase,
* patients who have experienced a greater than or equal to grade 3 allergic reaction to E. coli L-asparaginase and who have never received E. chrysanthemi L-asparaginase after the occurrence of this reaction,
* WBC count greater than 20 Gica/L, any of the following laboratory abnormalities if not due to hematologic malignancy (calculated creatinine clearance less than 50 mL/min,
* serum SGOT/AST or SGPT?ALT greater than 2.5 x upper limit of normal,
* serum total bilirubin greater than 2.0 mg/dL, except in the case of hemolytic anemia.
* Patients cannot have a history of greater than or equal to grade 2 pancreatitis,
* any history of allogeneic transplant,
* receiving steroid therapy with a dose greater than 20 mg/day,
* known HIV positive serology,
* active hepatitis B or C,
* any serious active disease or comorbid medical condition or psychiatric illness that would prevent the subject from signing the informed consent.
* Pregnant or lactating females or women of child bearing potential not willing to use an adequate method of birth control for the duration of the study are not eligible.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 6 months
  To determine the Maximum Tolerated Dose following one single dose of mPEG-r-Crisantaspase when administered in a population of patients with relapsed or refractory hematological malignancies, as measured by Dose Limiting Toxicities.

SECONDARY OUTCOMES:
Asparaginase Activity in serum | 6 months
  To determine the pharmacokinetic profile as assessed by measurement of serum L-asparaginase enzymatic activity following single and double mPEG-r-chrisantaspace doses.

CONTACTS AND LOCATIONS:
Overall Officials: Pr Gilles Salles, MD, Principal Investigator — Centre Hospitalier Lyon Sud -Chemin du Grand Revoyet; Xavier Thomas, MD, Study Director — Centre Hospitalier Lyon Sud - Chemin du Grand Revoyet
Locations (5):
- France (5):
  - Centre Henri Becquerel, Rouen, Cedex
  - Hôpital Henri Mondor, Créteil
  - Hôpitaux du CHU de Nantes, Nantes
  - Hospices Civils de Lyon, Pierre-Bénite
  - Institut Claudius Regaud, Toulouse